CLINICAL TRIAL: NCT04787497
Title: The Neuropsychological Effects of Extra-Virgin Olive Oil in People With Multiple Sclerosis
Brief Title: The Effect of Extra Virgin Olive Oil in People With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cyprus (Other)
Collaborators: World Olive Center for Health (Unknown); Ellis-Farm, Eliama Daily Value (Unknown)
Responsible Party: Principal Investigator, Maria Loizou, Clinical Psychology Doctorate Student, University of Cyprus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NEEVOO.MS
Record Dates: First submitted 2021-03-01; First posted 2021-03-08 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The Experimental Group will be receiving 50ml of freshly, cold-pressed, oleocanthal-rich Extra Virgin Olive Oil (EVOO) alongside their prescribed medical treatment. EVOO will be consumed on a daily basis for 12 months and all participants will undergo a neuropsychological assessment at baseline, 6 months and 12 months +/- 7 days after their first assessment or beginning of supplementation.
  Interventions: Dietary Supplement: High Phenolic Extra Virgin Olive Oil
- Control Group (No Intervention): The Control Group will be continuing their standard medical treatment without additional supplementation. The neuropsychological assessment will be conducted at baseline, 6 months and 12 months +/- 7 days after their first assessment.

INTERVENTIONS:
Dietary Supplement: High Phenolic Extra Virgin Olive Oil — Participants will be assigned in two groups: the Experimental Group (N= 20) will be receiving 50ml of freshly, cold-pressed, oleocanthal-rich Extra Virgin Olive Oil (EVOO) alongside their prescribed medical treatment, whereas the Control Group (N = 20) will be receiving their medical treatment as usual. The Experimental Group will be receiving the complementary treatment on a daily basis for 12 months and all participants will undergo a neuropsychological assessment at baseline, 6 months and 12 months +/- 7 days after their first assessment or beginning of treatment.
  Arms: Experimental Group

SUMMARY:
This is an open label feasibility trial to examine the effect of a complementary treatment with High Phenolic Extra Virgin Olive Oil (HPEVOO) on the cognitive and mental health of people with Multiple Sclerosis (MS), while receiving their standard medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MS
* Must be between 18 to 65 years of age
* Both males and females are eligible for participation
* Must have at least five years of education
* Must be fluent in Greek language

Exclusion Criteria:

* Other neurological, psychiatric or chronic condition
* Enrollment in other trials/drug studies
* Experiencing side effects from previous treatments
* Inadequate visual and auditory acuity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Symbol Digits Modalities Test (SDMT) | baseline, 6-months, 12-months
  Change will be assessed in the SDMT score (0-100 range), over three time points. Higher score indicates better processing speed.
California Verbal Learning Test-Second Edition (CVLT-II) | baseline, 6-months, 12-months
  Change will be assessed in the CVLT-II score (0-80 range), over three time points. Higher score indicates better auditory-verbal learning.
Brief Visuospatial Memory Test-Revised (BVMT-R) | baseline, 6-months, 12-months
  Change will be assessed in the BVMT-R score (0-36 range), over three time points. Higher score indicates better visuospatial memory.
Wisconsin Card Sorting Test (WCST) | baseline, 6-months, 12-months
  Change will be assessed in the WCST score over three time points. WCST examines attention, working memory and intellectual flexibility (0-64 score range). Higher scores represent worse performance.
Trail Making Test (TMT) | baseline, 6-months, 12-months
  Change will be assessed in the TMT scores over three time points. TMT examines attention, intellectual flexibility and inhibition. Longer time to completion indicates worse performance.
The Vocabulary and Block Design from the Wechsler Adult Intelligence Scale (WAIS) | baseline
  It will provide an estimated intelligence quotient (IQ) score
The Digit Span Test (DST) from WAIS | baseline, 6-months, 12-months
  Change will be assessed in the DST score over three time points. DST examines working memory, 0-48 score range, higher scores indicate better working memory function.
Word List Generation (WLG) Test | baseline, 6-months, 12-months
  Change will be assessed in the WLG score over three time points. WLG examines lexical fluency. The higher the number of words generated, the better is the performance.
Faux Pas Recognition (FPR) Test | baseline, 6-months, 12-months
  Change will be assessed in the FPR score over three time points. FPR examines social cognition. Four different vignettes will be used for every assessment (0-20 score range). Higher scores indicate better performance.
Hospital Anxiety and Depression Scale (HADS) | baseline, 6-months, 12-months
  Change will be assessed in the HADS scores over three time points. HADS examines anxiety, depression and psychological distress. Higher scores (0-42 range) indicate greater levels of anxiety and depression.
Health Status Questionnaire (SF-36) | baseline, 6-months, 12-months
  Change will be assessed in SF-36 scores over three time points. SF-36 consists of eight scales (0-100 score range each) that examine physical and mental health-related quality of life. The lower the score the more disability.
Modified Fatigue Impact Scale (MFIS) | baseline, 6-months, 12-months
  Change will be assessed in the MFIS score over three time points. MFIS examines how often fatigue interferes with daily activities. Higher scores (0-84 score range) indicate greater impact of fatigue on a person's activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Private medical office, Thessaloniki, Greece